CLINICAL TRIAL: NCT01840462
Title: A National, Multicenter, Non-interventional, Prospective, Longitudinal Study for Treatment With Botulinum Toxin A Injections in naïve and Pre-treated Patients Suffering From Cervical Dystonia (Dysport®)
Brief Title: Longitudinal Study for Treatment With Botulinum Toxin A Injections in naïve and Pre-treated Patients Suffering From Cervical Dystonia [CD-NIS-Longterm]
Acronym: CDNISLongterm
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-94-52120-165
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects naïve to botulinum toxin A (BoNT-A) treatment: Patients naïve to botulinum toxin A treatment
- Subjects pre-treated with botulinum toxin A (BoNT-A) injection: Patients pre-treated with botulinum toxin A for at least 2 years.
  4 injection cycles, each at 3 to 4 months intervals. Investigators follow their individual injection protocol for the treatment with BoNT-A (modalities of administration in accordance with local Summary of Product Characteristics).

SUMMARY:
The objective of this study is to investigate the efficacy of Dysport® in the treatment of cervical dystonia (CD) in a non-interventional long-term study in naïve and pre-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from cervical dystonia with rotational torticollis/-caput or laterocollis/-caput as the primary component
* Naïve to botulinum toxin A or pre-treated with botulinum toxin A on a regular basis for at least 2 years prior to inclusion and last injection with Dysport® and last injection between 3 and 6 months prior to inclusion
* With the intention to be treated with Dysport®

Exclusion Criteria:

* The subject has already been included in this study
* Participation in an interventional trial
* Suffering from anterocollis or retrocollis as primary component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from cervical dystonia
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Tsui scores | Baseline and 12 weeks post-injection Cycle 2
  The Tsui rating scale is a disease-specific score to evaluate the severity of CD taking the clinical signs of CD into account in a standardised manner.

SECONDARY OUTCOMES:
Change in Tsui scores | Baseline and 12 weeks post-injection Cycle 1
  The Tsui rating scale is a disease-specific score to evaluate the severity of CD taking the clinical signs of CD into account in a standardised manner.
Change in Tsui scores | Baseline and 12 weeks post-injection Cycle 3
  The Tsui rating scale is a disease-specific score to evaluate the severity of CD taking the clinical signs of CD into account in a standardised manner.
Change in Tsui scores | Baseline and 12 weeks post-injection Cycle 4
  The Tsui rating scale is a disease-specific score to evaluate the severity of CD taking the clinical signs of CD into account in a standardised manner.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Graz, Austria
- Wiesbaden, Germany